CLINICAL TRIAL: NCT02987530
Title: Phase III Multicenter Randomized Trial Evaluating in Patients At the Time of the Primary HIV-1 Infection, the Impact on the Viral Reservoir of a Combination Including Tenofovir/emtricitabine and Dolutegravir or Tenofovir/emtricitabine and Darunavir/cobicistat
Brief Title: National Multicenter Trial Evaluating Two Treatments in Patients with Primary Human Immunodeficiency Virus (HIV-1) Infection
Acronym: OPTIPRIM-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 169; 2016-001683-11 (EudraCT Number)
Record Dates: First submitted 2016-11-30; First posted 2016-12-09 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2019-08

CONDITIONS: HIV-1 Infection
Keywords: primary infection
MeSH Terms: interventions — dolutegravir; cobicistat mixture with darunavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dolutegravir + Emtricitabine/Tenofovir (Experimental): Patients will take Dolutegravir 50 mg (= Tivicay, 1 tablet per day) with Emtricitabine 200 mg / Ténofovir 245 mg (=Truvada, 1 tablet per day) for 48 weeks
  Interventions: Drug: Dolutegravir; Drug: Emtricitabine-Tenofovir
- Darunavir/Cobicistat + Emtricitabine/Ténofovir (Active Comparator): Patients will take Darunavir 800 mg / Cobicistat 150 mg (=Rezolsta, 1 tablet per day) + Emtricitabine 200 mg / Ténofovir 245 mg (=Truvada, 1 tablet per day) for 48 weeks
  Interventions: Drug: Darunavir-cobicistat; Drug: Emtricitabine-Tenofovir

INTERVENTIONS:
Drug: Dolutegravir — Oral use, 50mg/day
  Other Names: Tivicay
  Arms: Dolutegravir + Emtricitabine/Tenofovir
Drug: Darunavir-cobicistat — Oral use, 800-150mg/day
  Other Names: Rezolsta
  Arms: Darunavir/Cobicistat + Emtricitabine/Ténofovir
Drug: Emtricitabine-Tenofovir — Oral use, Emtricititabine : 200mg/day Ténofovir : 245mg
  Other Names: Truvada

SUMMARY:
The purpose of this study is to compare the impact of two combination of two tablets once daily: dolutegravir associated with emtricitabine / tenofovir versus darunavir / cobicistat associated with emtricitabine / tenofovir on DNA HIV measured in PBMC at 48 weeks in patients with primary HIV-1 infection.

DETAILED DESCRIPTION:
Phase III, randomized (1: 1), comparative, superiority, open-label, parallel assignment, national multicenter trial evaluating two treatments in patients with primary HIV-1 infection.

Comparison of the two combinations regarding:

* Viral reservoir at W48
* Early inhibition of viral replication,
* Plasmatic and cellular cumulative viremia at W48,
* Immune reconstitution with CD4, CD8 levels and CD4 / CD8 ratio,
* Activation parameters decrease,
* Adherence to treatments,
* Treatments tolerance,
* Adverse events,
* Quality of life (by self-administered questionnaires). Study of the pharmacokinetics / dynamics relationship of the decay of plasma, cellular and spermatic compartments' viral loads.

  50 participants per group will be enrolled in 40 sites in France. Co- inclusion in ANRS CO 06 PRIMO cohort will be offered

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at screening visit.
* Patients with primary HIV-1 infection: Any results achieved in the previous 10 days of inclusion visit will be taken into account. If the Enzyme Linked ImmunoSorbent Assay (ELISA) test result does not dissociate the signals antibodies and p24 antigen or in case of rapid test result :

  * Negative ELISA / rapid test and positive HIV-1 RNA confirmed by a second positive HIV-1 RNA.
  * Positive ELISA / rapid test and WB-HIV1 [0-5] band (s) or IB-HIV-1 [0-3] band(s) confirmed by a positive HIV-1 RNA.

If the ELISA test result dissociated p24 antigen and antibodies signals:

* ELISA Ac - / p24 - and positive HIV-1 RNA confirmed by a second positive HIV-1 RNA.
* ELISA Ac - / p24 + confirmed by a positive HIV-1 RNA.
* ELISA Ac + / p24 + or - and WB-HIV1 [0-5] band (s) or IB-HIV-1 [0-3] band(s) confirmed by a positive HIV-1 RNA.

  * Written informed consent signed by the person and the investigator no later than the day of the screening visit and before any exam performed in the trial (article L1122-1-1 Public Health Code).
  * Affiliate or beneficiary of a social security system (Article L1121-11 of the Public Health Code) (the State Medical Aid or AME is not a social security system).
  * Patients followed in selected centers, accepting additional constraints and having signed a consent, will participate to virological, immunological and pharmacological sub-studies.
  * Patient agreeing to participate in the trial for 1 year according to the defined terms.

Exclusion Criteria:

* Any antiretroviral treatment (for Pre-Exposure Prohylaxis or Post-exposure prophylaxis) during the 4 weeks preceding inclusion.
* Associated pathology with urgent care needed.
* Prothrombin Ratio < 50%.
* Creatinine clearance < 70 mL / min (Cockroft).
* aspartate transaminase (AST), alanine transaminase (ALT), or bilirubin (total and conjugated) ≥ 10 times the upper limit of normal.
* Patient with isolated HIV-2 viral strain.
* Women of childbearing potential without effective contraception method (see appendix A6).
* Pregnant or breastfeeding women.
* Person under legal guardianship or deprived of liberty by a judicial or administrative decision.
* Patient participating in another research evaluating other treatments with an exclusion period ongoing at the screening visit.
* Planned absence which could prevent optimal trial participation (vacation abroad, moving, imminent job change ...).
* Co-administration of prohibited treatments (see § 9.5).
* History or presence of allergy to the study drugs or their components;
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects with severe hepatic impairment (Class C) as determined by Child-Pugh classification.
* Any symptoms or laboratory values suggesting a systemic disorder (renal, hepatic, cardiovascular, pulmonary) or other medical conditions that could interfere with the interpretation of trial results or compromise the health of patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
HIV-DNA levels in the peripheral blood mononuclear cell (PBMC) at week 48 | week 48

SECONDARY OUTCOMES:
Cumulative cellular viremia up to week 48 | week 48
Cumulative plasmatic viremia (HIV-1 RNA) at week 48 | week 48
Cumulative plasmatic viremia using the values obtained by ultrasensitive quantification for all HIV-1-RNA values < 50 copies / mL. | week 48
Levels of HIV-1 RNA in plasma at week 2, week 4, week 8, week 12, week 24, week 36, week 48 and changes between week 0 and week 48 | week 2, week 4, week 8, week 12, week 24, week 36, week 48
Percentage of patients with HIV-1 RNA <50 copies / mL at week 2, week 4, week 8, week 12, week 24, week 36, week 48 | week 2, week 4, week 8, week 12, week 24, week 36, week 48
Proportion of patients with HIV-1-RNA plasma below the ultrasensitive technique quantification threshold at week 2, week 4, week 8, week 12, week 24, week 36 and week 48 | week 2, week 4, week 8, week 12, week 24, week 36 and week 48
Total DNA-HIV levels measured in PBMC at week 2, week 4, week 8, week 12, week 24, week 36 and week 48 | week 2, week 4, week 8, week 12, week 24, week 36 and week 48
Total DNA-HIV levels measured in PBMC: changes between week 0 and week 48. | between week 0 and week 48
CD4 and CD8 counts and percentage at week 2, week 4, week 8, week 12, week 24, week 36, week 48. | week 2, week 4, week 8, week 12, week 24, week 36, week 48
CD4 and CD8 counts and percentage changes between week 0 and week 48. | between week 0 and week 48.
CD4/CD8 ratio at week 2, week 4, week 8, week 12, week 24, week 36, week 48. | week 2, week 4, week 8, week 12, week 24, week 36, week 48
CD4/CD8 ratio changes between week 0 and week 48. | between week 0 and week 48.
Pharmacokinetic: mean concentrations between week 0 and week 48 will be linked to plasma RNA-VIH and DNA-VIH decrease. | between week 0 and week 48
Pharmacokinetic: cumulative AUC between week 0 and week 48 will be linked to plasma RNA-VIH and DNA-VIH decrease. | between week 0 and week 48
Trial treatments tolerance using self-administered questionnaires of symptoms experienced. | week 0, week 4, week 8, week 12, week 24, week 36 and week 48
Reported quality of life using self-administered questionnaire (PROQOL-HIV questionnaire). | between week 0 and week 48
Number, nature and time of occurrence of stage 3 or 4 clinical and biological adverse events (using ANRS scale to grade severity of adverse events in adults). | between week 0 and week 48
HIV infection progression defined by occurrence of B or C stage clinical events or death between week 0 and week 48 | between week 0 and week 48
Evolution of Metabolic disorders assessed by measurement of cholesterol, triglycerides, blood glucose and lipase | between week 0 and week 48
Evolution of Renal function assessed by urea and serum creatinine. | between week 0 and week 48
Adherence to treatments using self-administered questionnaires | week 4, week 8, week 12, week 24, week 36 and week 48
Adherence to treatments using pills' counts by local pharmacist | week 4, week 8, week 12, week 24 and week 36
Adherence to treatments using MEMS (Medical Event Monitoring System) data collected during the first 3 months | between week 0 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Chéret, MD, PhD, Principal Investigator — Hôpital Bicêtre
Locations (1):
- Hopital Bicetre, All the Regions of the Country (40 Centers), France

IPD SHARING:
Plan to Share IPD: No